CLINICAL TRIAL: NCT01718431
Title: Prebiotics as Means to Modulate Colonic Events, With the Purpose to Increase Beneficial Effects on Metabolism, Satiety and Cognition.
Brief Title: Prebiotics as a Means to Modulate Gut Fermentation, Metabolism, Appetite and Cognition
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Elin Johansson, MSc, postgraduate student, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Dnr2010/457 - 3day
Record Dates: First submitted 2012-10-09; First posted 2012-10-31 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- indigestible carbohydrates (Experimental): test meal: indigestible carbohydrates
  Interventions: Other: test meal
- reference (Experimental): reference meal: no indigestible carbohydrates
  Interventions: Other: reference meal

INTERVENTIONS:
Other: test meal
  Arms: indigestible carbohydrates
Other: reference meal
  Arms: reference

SUMMARY:
This study aims at investigating the impact of colonic fermentation of intrinsic indigestible carbohydrates in cereal whole kernels after three days consumption, on metabolic variables and cognition. The study is performed in healthy, normal to slightly over-weight test subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI 19-28 kg/m2

Exclusion Criteria:

* gastrointestinal diseases
* metabolic disorders
* tobacco/snuff user
* antibiotic/probiotic treatment

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of the test meal | Post-prandially after breakfast, 0-150 min
  The differences in AUC between different risk markers, assessed in plasma or serum,after intake of the test meal in comparison to the reference meal is measured. Example of variables measured are glucose, insulin, appetite hormones, inflammatory markers, markers of colonic fermentation.

SECONDARY OUTCOMES:
Cognitive performance | Post-prandially after breakfast, 0-210 min
  The cognitive performance of the test subjects is measured to investigate work memory and specific attention.
Subjective satiety | post-prandially after breakfast, 0-150 min
  The subjective sensation of satiety, hunger and desire to eat is measured using a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Nilsson, PhD, Principal Investigator — Lund University
Locations (1):
- Applied Nutrition and Food Chemistry, Lund University, Lund, Sweden

REFERENCES:
- [Derived] Nilsson AC, Johansson-Boll EV, Bjorck IM. Increased gut hormones and insulin sensitivity index following a 3-d intervention with a barley kernel-based product: a randomised cross-over study in healthy middle-aged subjects. Br J Nutr. 2015 Sep 28;114(6):899-907. doi: 10.1017/S0007114515002524. Epub 2015 Aug 11. PMID 26259632